CLINICAL TRIAL: NCT04806204
Title: Effect of Music Therapy on Pain, Anxiety and Vital Signs Before and During Coronary Angiography
Brief Title: Music Therapy in Coronary Angiography
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: BAIBU-ANG-ELF
Record Dates: First submitted 2021-01-27; First posted 2021-03-19 (Actual); Last update posted 2021-09-30 (Actual); Status verified 2021-09

CONDITIONS: Nursing Caries; Complementary Therapies; Cardiology
Keywords: Coronary Angiography; Music Therapy; Vital Signs; Anxiety
MeSH Terms: conditions — Anxiety Disorders | interventions — Music Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- music therapy before the angiography (Experimental): Patients in the Intervention 1 group will be offered Turkish Folk, Classical, Turkish Art and Sufi Music as an option, and the music preferred by the patients will be played with headphones for 15-20 minutes before the CAG procedure. Since individuals are in the CAG unit collectively before the procedure, headphones will be used in order not to disturb other individuals. After the interviews, musical types will be arranged as instrumental, non-verbal, at 70 decibels, approximately 60 metronome per minute, in terms of rhythm and duration, and will be played according to the individual's choice. Instrumental works will be uploaded to the portable MP3 player provided by the researchers.
  Interventions: Other: music therapy
- music therapy during the angiography (Experimental): Patients in the Intervention 2 group will be offered Turkish Folk, Classical, Turkish Art and Sufi Music as an option, and the music preferred by the patients will be played through a speaker that will be placed in the CAG hall during the CAG procedure. After the interviews, musical types will be arranged as instrumental, non-verbal, 75 decibels, approximately 60 metronome per minute, in terms of rhythm and duration, and will be played according to the individual's choice.
  Interventions: Other: music therapy
- control group (No Intervention): After the polyclinic controls of the patients, on the day of the CAG procedure, data collection forms will be applied in the CAG unit 30 minutes before the procedure. Routine care will be applied to patients in this group and music therapy will not be applied. The physiological parameters of the patient will be measured by the clinical nurse 15 minutes after the procedure, and data collection forms will be applied again 20 minutes later.

INTERVENTIONS:
Other: music therapy — Music therapy will be applied to one group before angiography and to the other group during angiography. Patients who will listen to music before angiography will be offered Turkish Folk, Classical, Turkish Art and Sufi Music as an option, and the music preferred by the patients will be played with headphones for 15-20 minutes. Patients who will listen to music during angiography will be offered Turkish Folk, Classical, Turkish Art and Sufi Music as an option, and the music preferred by the patients will be played through a speaker that will be placed in the angiography hall during the angiography procedure.
  Arms: music therapy before the angiography; music therapy during the angiography

SUMMARY:
Aim: This study was planned as randomized controlled to determine the effect of music therapy applied before and during angiography on pain, anxiety and physiological parameters after angiography.

The study was planned as a pre-test, post-test design, single center, randomized controlled experimental study.The study is planned to be conducted in the coronary angiography (CAG) unit of a university hospital between January 2021 and December 2021., the study sample will be composed of a total of 102 individuals, 34 in each group (intervention 1 group listening to music before the procedure = 34, intervention 2 group listening to music during the procedure = 34, control group = 34).Data in the research; The Introductory Form will be collected using the State-Trait Anxiety Scale, Vital Signs Follow-up Form and Visual Pain Scale (VAS).Patients in the Intervention 1 group will be offered Turkish Folk, Classical, Turkish Art and Sufi Music as an option, and the music preferred by the patients will be played with headphones for 15-20 minutes before the CAG procedure.Patients in the Intervention 2 group will be offered Turkish Folk, Classical, Turkish Art and Sufi Music as an option, and the music preferred by the patients will be played through a speaker that will be placed in the angiography hall during the CAG procedure. Routine care will be applied to patients in this group and music therapy will not be applied.

DETAILED DESCRIPTION:
It is predicted that music therapy will be beneficial before and during angiography in order to prevent complications, reduce anxiety and pain, and provide patient comfort and satisfaction. This study was planned as randomized controlled to determine the effect of music therapy applied before and during angiography on pain, anxiety and physiological parameters after angiography.

Material - Method Research design: The study was planned as a pre-test, post-test design, single center, randomized controlled experimental study.

Place and Time of the Study: The study is planned to be conducted in the coronary angiography(CAG) unit of a university hospital between January 2021 and December 2021.

Population and sampling: The population of the study consists of patients who will undergoing CAG between January 2021 and December 2021. No special method is used for sample selection, individuals who are treated on the specified dates, who meet the inclusion criteria and who volunteer to participate in the study will be included in the sample. Power analysis will be done to determine the sample size. The sample of the study will be composed of individuals who meet the inclusion criteria of the study within the time that the study is planned. As a result of the literature review, the number of samples for each group was found to be 28 at a significance level of α = 0.05 and a power of 80% in randomized controlled studies with CAG. However, considering that there may be losses in the implementation phase of the study, provided that the individuals who will be treated with CAG are included, 20% more of these numbers in each group will be included in the study. Thus, the study sample will be composed of a total of 102 individuals, 34 in each group (intervention 1 group listening to music before the procedure = 34, intervention 2 group listening to music during the procedure = 34, control group = 34). In addition, while the application of the study continues, the data obtained will be transferred to the computer program and it will be evaluated whether the sufficient sample number has been reached by power analysis.

Data Collection Tools Data in the research; The Introductory Form will be collected using the State-Trait Anxiety Scale, Vital Signs Follow-up Form and Visual Pain Scale.

Patient Information Form This form consists of 17 questions in order to determine the personal information of the patients (age, gender, occupation, educational status, marital status, people living with them, income level, smoking-alcohol use, family angiography history, social security, etc.).

State-Trait Anxiety Scale The original of this scale was developed by Spielberger et al. In 1970 to determine the level of anxiety. It consists of two parts as "State and Trait Anxiety Scale".

* State Anxiety Scale: It is a 4-point Likert type scale consisting of 20 questions aiming to measure how individuals feel at the moment. The scores obtained from the scale vary between 20 and 80, and a high score indicates that anxiety is high, and a low score indicates that anxiety level is low. The adaptation to the Turkish form was made by Öner and Le Compte. In the state anxiety scale; There are two types of expressions: direct expressions expressing negative feelings and inverted statements expressing positive feelings. The expressions to be scored in reverse in the State Anxiety Scale are items 1, 2, 5, 8, 10, 11, 15, 16, 19 and 20. While these items are scored, those with 1 weight value are converted to 4, and those with 4 weight values are converted into 1 and the score is calculated. A total score of 0-19 from the scale indicates that there is no anxiety, the total score between 20-39 indicates mild, the total score between 40-59 indicates moderate, and the total score between 60-79 indicates severe anxiety, while 60 points above indicate the need for professional help. Test-retest reliability of the scale was found between 0.16 and 0.54.
* Trait Anxiety Scale: Indicates how the person feels regardless of the situation and conditions. Scores from each scale range between 20 and 80. A high score means high, and a low score means a low level of anxiety. The same is true when interpreting the scores in order of percentage. That is, a low percentage (1, 5, 10) shows that anxiety is low. The average score level determined in the applications varies between 36 and 41. 0-30 indicates low anxiety, 31-49 indicates moderate anxiety, and 50 and above indicate high anxiety. The expressions with reverse scoring on the Spielberg Trait Anxiety Scale are 1, 6, 7, 10, 13, 16, 19. Test-retest reliability was found between 0.73 and 0.86.

Vital Signs Follow-up Form This form; It was prepared with the aim of recording body temperature, pulse, blood pressure, oxygen saturation and respiratory values from vital signs of the individual measured before and after the procedure. The vital signs of the patients measured by the clinical nurses before and after the procedure and recorded on the nurse observation form will be recorded in the vital signs follow-up form by the investigators.

Visual Pain Scale Visual analog scale was used to evaluate the pain. It consists of a straight line with endpoints defining the extremes such as "no pain" and "pain as bad as possible". The patient is asked to mark the pain level on the line between the two end points. This tool was first used in psychology by Freyd in 1923. Kersten et al. Proved in their study that VAS is a valid tool for pain assessment. This results in accordance with Unsal and Ergül vase 2.9% rate in their study has determined that it is being used in studies in Turkey. The horizontal form of VAS will be used in the assessment of pain in our study.

Data Collection Individuals meeting the inclusion criteria in data collection will be randomized into 3 groups. Individuals who meet the inclusion criteria in the study will be randomized in a computer program and divided into intervention group 1, intervention group 2 and control group. Individuals undergoing elective angiography will be included in the groups according to their arrival order. In the randomization table, the first column represents the "intervention 1 group", the second column represents the "intervention 2 group", and the third column represents the "control group". Patients who meet the inclusion criteria will be included in the group in which column they are included in the order of arrival.

Intervention 1 Group After the polyclinic controls of the patients, on the day of the CAG procedure, data collection forms will be applied in the CAG unit 30 minutes before the procedure. Patients in the Intervention 1 group will be offered Turkish Folk, Classical, Turkish Art and Sufi Music as an option, and the music preferred by the patients will be played with headphones for 15-20 minutes before the CAG procedure. Since individuals are in the CAG unit collectively before the procedure, headphones will be used in order not to disturb other individuals. In determining the music to be played, literature was searched and expert opinion was obtained from the academicians of Fine Arts Education Department Music Department. After the interviews, musical types will be arranged as instrumental, non-verbal, at 70 decibels, approximately 60 metronome per minute, in terms of rhythm and duration, and will be played according to the individual's choice. Instrumental works will be uploaded to the portable MP3 player provided by the researchers. The patients in the Intervention 1 group will be introduced to the MP3 player before the procedure and how they should use it and the questions of the patients will be answered. After the patients who are taken to the CAG unit for the CAG procedure are prepared for the operation, the patients will be told to imagine that the outcome of the procedure will be positive, headphones will be worn and music therapy will be started. In addition, patients will be informed that they can interfere with the sound of the music, turn the sound on and off, stop the music and start listening again if they wish. The physiological parameters of the patient will be measured by the clinical nurse 15 minutes after the procedure, and data collection forms will be applied again after 20 minutes.

Intervention 2 Group After the polyclinic controls of the patients, on the day of the angiography procedure, data collection forms will be applied in the angiography unit 30 minutes before the procedure. Patients in the Intervention 2 group will be offered Turkish Folk, Classical, Turkish Art and Sufi Music as an option, and the music preferred by the patients will be played through a speaker that will be placed in the CAG hall during the CAG procedure. In determining the music to be played, literature was searched and expert opinion was obtained from the academicians of Fine Arts Education Department Music Department. After the interviews, musical types will be arranged as instrumental, non-verbal, 75 decibels, approximately 60 metronome per minute, in terms of rhythm and duration, and will be played according to the individual's choice. The physiological parameters of the patient will be measured by the clinical nurse 15 minutes after the procedure, and data collection forms will be applied again after 20 minutes.

Control Group After the polyclinic controls of the patients, on the day of the aCAG procedure, data collection forms will be applied in the angiography unit 30 minutes before the procedure. Routine care will be applied to patients in this group and music therapy will not be applied. The physiological parameters of the patient will be measured by the clinical nurse 15 minutes after the procedure, and data collection forms will be applied again 20 minutes later.

Ethical considerations: Ethical approval will be obtained from the "Bolu Abant İzzet Baysal University Clinical Research Ethics Committee" in order to conduct the study. Institutional permission will be obtained from "Izzet Baysal Training and Research Hospital where the study will be conducted. In addition, before starting the application, written consent will be obtained by the researcher explaining the purpose of the study to those who meet the inclusion criteria of the study.

Data analysis: In evaluating the data, the significance level was taken as p <0.05, and the data will be analyzed using the SPSS (25.00) program. In the evaluation of the data, besides descriptive statistical methods (frequency, percentage and average), Independent Samples Unrelated samples t test will be used for intergroup comparisons of parameters showing normal distribution, and related samples t test will be used for intragroup comparisons. In the intergroup comparisons of non-normally distributed parameters, Kruskall Wallis will be used to determine the significant difference of variables with more than three subcategories, the Mann Whitney U will be used to determine the group that causes the difference, and the Wilcoxon signed rank test (for the same group data) will be used for intragroup comparisons of non-normally distributed parameters.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Can speak and understand Turkish
* No hearing problems
* Oriented to place and time
* Have no psychiatric illness
* Sedative or analgesic medication within the last 24 hours
* where the intervention will be made in the ral zone
* The first time angiography procedure will be applied
* Individuals who are volunteers will be included in the study.

Exclusion Criteria:

* Under the age of 18
* Do not speak Turkish
* Have a hearing problem
* Without a place and time orientation
* Have any psychiatric illness
* Using sedative or analgesic drugs in the last 24 hours
* To be intervened outside the femoral area
* Previous angiography procedure
* Non-volunteer individuals will not be included in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2021-01-27 (Actual); Primary Completion 2021-12-27 (Estimated); Study Completion 2021-12-27 (Estimated)

PRIMARY OUTCOMES:
Means of subjective anxiety scores | up to 20 minutes post-angiography
  State-Trait Anxiety Scale is used to measure subjective anxiety. The original of this scale was developed by Spielberger et al. In 1970 to determine the level of anxiety. It consists of two parts as "State and Trait Anxiety Scale". State Anxiety Scale is a 4-point Likert type scale consisting of 20 questions aiming to measure how individuals feel at the moment. The scores obtained from the scale vary between 20 and 80, and a high score indicates that anxiety is high, and a low score indicates that anxiety level is low.
  The 20-item trait anxiety inventory shows the general feelings of the person under the situation and conditions.Scores from each scale range between 20 and 80. A high score means high, and a low score means a low level of anxiety.
Means of subjective pain scores | up to 15 minutes post-angiography
  The visual pain scale will be used to assess the patient's subjective pain. The patient will be asked to score his pain on the scale from 0 to 10. Average pain scores will be calculated for pain assessment.
Means of body temperature (0C) | up to 15 minutes post-angiography
  It will be measured by the clinical nurse using an infrared thermometer.
Means of systolic blood pressure (mmHg) | up to 15 minutes post-angiography
  The measurement on the arm, which is not operated with a digital blood pressure meter, will be made by the clinical nurse.
Means of diastolic blood pressure (mmHg) | up to 15 minutes post-angiography
  The measurement on the arm, which is not operated with a digital blood pressure meter, will be made by the clinical nurse.
Means of heart rate (/minutes) | up to 15 minutes post-angiography
  It will be measured by the clinical nurse with a pulse oximeter in the unprocessed arm.
Means of respiratory rate (/minutes) | up to 15 minutes post-angiography
  It will be counted by the clinical nurse by monitoring chest movements for one minute.
Means of oxygen saturation (%) | up to 15 minutes post-angiography
  It will be measured by the clinical nurse with a pulse oximeter in the unprocessed arm.

CONTACTS AND LOCATIONS:
Overall Officials: Saadet Can Cicek, Dr., Principal Investigator — Bolu Abant Izzet Baysal University, Health Sciences Faculty
Locations (1):
- Bolu Abant Izzet Baysal University Izzet Baysal Training and Research Hospital, Bolu, Center, Turkey (Türkiye)